CLINICAL TRIAL: NCT02828007
Title: Changes in Lung Ventilation With Different Modes of Non-invasive Ventilation in Healthy Subjects
Brief Title: EIT Study With Healthy Patients
Acronym: EIT Step 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: B&D Electromedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 185543
Record Dates: First submitted 2016-02-12; First posted 2016-07-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Participants
Keywords: EIT; NIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment/Intervention (Experimental): Each patient will be using Non Invasive Ventilation (NIV) and will use it on each possible ventilation mode in a random order with a 10 minutes washout period between modes.
  Interventions: Device: NIV Group

INTERVENTIONS:
Device: NIV Group — Each patient will be using Non Invasive Ventilation (NIV) and will use it on each possible ventilation mode in a random order with a 10 minutes washout period between modes.

SUMMARY:
Patients with severe respiratory diseases such as chronic obstructive pulmonary disease (COPD) or obesity-hypoventilation syndrome (OHS) can benefit from having non-invasive ventilation (NIV). Non-invasive ventilation consists of a machine (ventilator) that is blowing air through a mask. NIV provides patients with a bigger expansion of their lung when they are breathing. This better expansion helps patients to have more oxygen and less waste gas (or carbon dioxide) in their body.

These improvements enhance survival and quality of life. In order to provide appropriate ventilation for each patient, the ventilator can generate different types of blowing:

* Continuous positive airway pressure (CPAP) which delivers a constant pressure to the mask
* Pressure support ventilation (PSV) which delivers a constant pressure to the mask and, on top of that, delivers more pressure when the patient begins to breathe in.
* Pressure control ventilation (PCV), which is similar to PSV, but use a fixed time to generate the flow when the patient begins to breathe in.

These different types of blowing have consequences on patient comfort as well as on the improvement of their ventilation.

To assess the improvement of the ventilation, the investigators currently use blood tests, however, these reflect overall output and may miss more subtle changes in breathing that could affect how patients feel.

Electrical impedance tomography (EIT) is a new technology that involves wearing a belt of sensors around the chest that provides information on how well the lungs are being filled with air by the ventilator. It allows a non-invasive assessment of the effect of NIV onto lung ventilation in real-time.

The investigators hope to use the EIT technology to assess in real-time patients lung ventilation when they are using the NIV. The investigators hope that EIT will provide them with information on which type of blowing is more effective and more comfortable than the others.

DETAILED DESCRIPTION:
Chronic lung disease can sometimes progress to the extent that patients can no longer clear the waste gas from their blood. Treatment can be offered with a mask and machine (ventilator) that helps people breathe and aims to improve their lung condition. It is common for people's lungs to be affected variably, i.e. left more than right or top of lung more than bases of lungs. The way in which the ventilator is set may affect how well the machine deals with these differences. If the lung is better ventilator patients may find the machine more comfortable and it may be more effective.

Electrical impedance tomography (EIT) is a new technology that involves wearing a belt of sensors around the chest that provides information on how well the lungs are being filled with air by the ventilator. It allows the assessment of these differences, which previously required the use of invasive equipment to obtain.

Optimising ventilator settings in the administration of non-invasive ventilation (NIV) can be improved with the addition of individual physiological data. This approach is limited due to the invasive techniques required to obtain this information, often leading to less ideal NIV settings promoting patient-ventilator asynchrony. It has been recently demonstrated by our group that all patients established on domiciliary NIV have a degree of patient-ventilator asynchrony and that the commonest type of asynchrony are triggering issues. Triggering asynchrony is promoted by mismatch between a patient's intrinsic positive end-expiratory pressure (iPEEP) and applied expiratory positive airway pressure (EPAP) with these ineffective efforts contributing to an increased work of breathing and patient discomfort. Previous strategies used to optimise patient triggering have involved the placement of oesophageal catheters in order to measure neural respiratory drive (NRD) to the diaphragm by electromyography (EMG) but again this process is invasive and often poorly tolerated. Electrical Impedance Tomography (EIT) is a non-invasive, bedside monitoring technique that provides semi-continuous, real-time information about the regional distribution of the changes in electrical resistivity of the lung tissue due to variations in ventilation in relation to a reference state.

Information is gained by repeatedly injecting small alternating electric currents (usually 5 mA) at high frequency of 50 - 80 kHz through a system of skin electrodes (usually 16) applied circumferentially around the thorax in a single plane between the 4th and 6th intercostal space. While an adjacent pair of electrodes 'injects' the current ('adjacent drive configuration'), all the remaining adjacent passive electrode pairs measure the differences in electric potential. A resistivity (impedance) image is reconstructed from this data by a mathematical algorithm using a two dimensional model and a simplified shape to represent the thoracic cross-section.

The resulting image possesses a high temporal and functional resolution making it possible to monitor dynamic physiological phenomena (e.g. delay in regional inflation or recruitment) on a breath by breath basis. It is important to realize that the EIT images are based on image reconstruction techniques that require at least one measurement on a well-defined reference state. All quantitative data are related to this reference and can only indirectly quantify (relative) changes in local lung impedance (but not absolute).

EIT can be used in mechanically ventilated patients to assess recruitment and to optimise ventilator settings to reduce risk of iatrogenic ventilator associated lung injury.

To date, EIT has only been validated in patient invasively ventilated or during self-ventilation.

The investigators hope to use the EIT technology to assess patients breathing using different ventilator modes in order to see if one is more effective and or more comfortable than the others. The investigators can use this information to help them set ventilators for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any underlying lung disease
* FEV1/FVC > 70%

Exclusion Criteria:

* Pregnancy
* Aged <18, >80
* Significant physical or psychiatric comorbidity
* that would prevent compliance with trial protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Characteristics seen during ventilation in different modes of ventilation | 1 day

SECONDARY OUTCOMES:
Correlation between tidal volume assessed by EIT | 1 day
Correlation between tidal volume assessed by NIV software | 1 day
Detection of patient ventilator asynchrony using physiological measurements | 1 day
Measurements of Neural Respiratory Drive using parasternal EMG | 1 day
Patient Comfort using Visual Analogue Scale | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, Study Chair — GSTT
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No